CLINICAL TRIAL: NCT06024382
Title: The Effect of Low-level Laser Therapy on Functional Treatment of Skeletal Class II Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nada Gaballah, teaching assistant, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dentist.1995
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Class II Malocclusion
Keywords: twin block , functional appliance , low level laser , photobiomodulation
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- twin block (Experimental): group treated with twin block only
  Interventions: Other: twin block
- twin block combined with low level laser (Experimental): group treated with twin block combined with low level laser therapy
  Interventions: Other: twin block combined with low level laser

INTERVENTIONS:
Other: twin block — 2 parallel groups one is treated with twin block and the other is treated with twin block combined with low level laser therapy
  Arms: twin block
Other: twin block combined with low level laser — 2 parallel groups one is treated with twin block and the other is treated with twin block combined with low level laser therapy
  Arms: twin block combined with low level laser

SUMMARY:
this is a controlled clinical trial with 2 groups of patients of class II skeletal discrepancy due to mandibular retrusion one group is treated with twin block functional appliance and the other with twin block combined with low level laser therapy ,the study aims to detect the effect of low level laser on the skeletal outcomes , dentoalveolar outcomes, rate of correction and pain during treatment

ELIGIBILITY:
Inclusion Criteria:

* Age (early permanent dentition)
* Cervical maturation stage CS 3-4
* Skeletal class II due to mandibular retrusion.
* Overjet more than 4mm.

Exclusion Criteria:

* Cleft lip or palate.
* Systemic diseases.
* Previous orthodontic treatment or abnormal habits.
* Congenital craniofacial deformity.
* poor oral hygiene

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
treatment time | 8 months
  comparison of treatment between the 2 different groups

SECONDARY OUTCOMES:
cephalometric measurements | 8 months
  digital tracing of pre and post treatment cephalograms of both groups and comparison of linear and angular measurements
study cast analysis | 8 months
  cast analysis of both groups measuring arch perimeter , intercanine wisth and intermolar width
the short form McGill pain questionnaire | 1 month
  comparison of questionnaire results between the 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No